CLINICAL TRIAL: NCT05837065
Title: Development and Validation of Novel Models Including Tumor Micronecrosis for Predicting the Postoperative Survival of Patients With Hepatocellular Carcinoma
Brief Title: Prognostic Models for HCC Based on Tumor Micronecrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Director, Zhejiang University
Other Study IDs: PMforHCC
Record Dates: First submitted 2023-04-17; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Tumor micronecrosis; Nomogram
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training cohort: HCC patients receiving curative hepatic resection
  Interventions: Other: observing whether HCC patients having tumor micronecrosis
- validation cohort: HCC patients receiving curative hepatic resection
  Interventions: Other: observing whether HCC patients having tumor micronecrosis

INTERVENTIONS:
Other: observing whether HCC patients having tumor micronecrosis — whether HCC patients having tumor micronecrosis or not

SUMMARY:
The heterogeneity of hepatocellular carcinoma (HCC) leads to the unsatisfying predicting performance of current staging systems. HCC patients with pathological tumor micronecrosis have immunosuppressive microenvironment. We aimed to develop novel prognostic models by integrating micronecrosis to more precisely predict the survival of HCC patients after hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically diagnosed as HCC;
2. curative hepatectomy with R0 resection;
3. conserved liver function with Child Pugh class A or B

Exclusion Criteria:

1. with macrovascular invasion or extrahepatic metastasis;
2. receiving other anti-tumor treatments such as TACE or systemic drugs;
3. with other primary cancers;
4. incomplete follow-up data;
5. without sufficient formalin-fixed, paraffin-embedded (FFPE) specimens for micronecrosis evaluation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study enrolled HCC patients receiving curative hepatectomy in the First Affiliated Hospital, Zhejiang University School of Medicine (FAHZU) (n = 765)
Sampling Method: Non-Probability Sample
Enrollment: 765 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
the Harrell concordance index (C-index) | Up to 5 years

SECONDARY OUTCOMES:
the time-dependent area under the receiver operating characteristic curve(tdAUROC) | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No